CLINICAL TRIAL: NCT02928250
Title: Role of Carnosine as an Adjuvant Therapy for Diabetic Nephropathy in Pediatrics With Type 1 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Nancy Samir Elbarbary, Ass.Prof.Nancy Samir Elbarbary, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Ain Shams University 1361
Record Dates: First submitted 2016-10-07; First posted 2016-10-10 (Estimated); Last update posted 2016-10-10 (Estimated); Status verified 2016-10

CONDITIONS: Type 1 Diabetes; Oxidative Stress; Carnosine; Diabetic Nephropathy
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetic Nephropathies | interventions — Carnosine

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- Carnosine oral daily (Active Comparator): Intervention group included pediatric patients with diabetic nephropathy receiving oral carnosine daily.
  Interventions: Dietary Supplement: Carnosine
- Second arm received placebo oral daily (Placebo Comparator): Placebo group or control patients received placebo that were similar in appearance to carnosine capsules and the administered dose was as the same schedule as carnosine.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Carnosine — Patients in intervention group received carnosine capsules orally daily
  Arms: Carnosine oral daily
Dietary Supplement: Placebo — Patients in placebo group received placebo that were similar in appearance to carnosine capsules and the administered dose was as the same schedule as carnosine.
  Arms: Second arm received placebo oral daily

SUMMARY:
Carnosine, a naturally-occurring dipeptide (β-alanyl-L-histidine) first described in 1900 by Gulewitsch and Amiradzibi, is found predominantly in post-mitotic tissues (e.g. brain and innervated muscle) of vertebrates . Carnosine is claimed to decrease oxygen free-radical mediated damage to cellular macromolecules either by chelating divalent cations or scavenging hydroxy radicals with its imidazole moiety. Free-radical damage is not the only process to affect the structure of proteins and nucleic acids.

To the best of our knowledge, no previous study assessed the role of carnosine in diabetes associated complications in particular diabetic nephropathy and there is insufficient evidence to recommend its supplementation in those patients. Therefore, this study was undertaken to investigate the role of carnosine as an adjuvant therapy for diabetic nephropathy in children and adolescents with type 1 diabetes and assess its relation to microalbuminuria, tubulointerstitial damage marker, glycemic control and oxidative stress.

ELIGIBILITY:
Inclusion Criteria:

* patients with type 1 diabetes.
* have diabetic nephropathy (≤18 years with at least 5 years disease duration )

Exclusion Criteria:

* any clinical evidence of infection, renal impairment due to causes other than diabetes, elevated liver enzymes, hypertension, neoplasm, hypersensitivity to carnosine, and taking any vitamins or food supplements one month before study or participation in a previous investigational drug study within the 30 days preceding screening.

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 90 (Actual)
Dates: Start 2015-08; Primary Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
effect on on urinary albumin excretion (UAE) | three months

SECONDARY OUTCOMES:
effect on alpha 1 microglobulin(A1M)) | three months
total antioxidant capacity (TAC), malondialdhyde (MDA). | three months